CLINICAL TRIAL: NCT01499862
Title: Discriminatory Neurosensory Stimulation Neurological H5394-11417-15
Brief Title: Mobility Training Using a Bionic Knee Orthosis in Patients Chronic Post-Stroke: A Case Series
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tibion Bionics, Inc. (Industry)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP 0003
Record Dates: First submitted 2011-12-20; First posted 2011-12-26 (Estimated); Results first posted 2013-08-02 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2013-06

CONDITIONS: Stroke
Keywords: Stroke; Tibion; Bionics; Rehab; Therapy; Robotics; Intention
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tibion Arm (Experimental): Arm of the study in which enrolled post-stroke subjects undergo rehabilitative therapy with the Tibion Bionic Leg.
  Interventions: Device: Tibion Bionic Leg

INTERVENTIONS:
Device: Tibion Bionic Leg — A programmable, carbon-fiber robotic leg orthosis (Tibion Bionic Leg, Tibion Corporation, Sunnyvale, CA) was used during therapy to actively supplement concentric and eccentric quadriceps function on the participant's impaired side. The device uses internal sensors at the foot and knee joint to detect intention of movement and, once a variable force threshold is passed, the devices provides appropriate assistive and resistive adjustments.

SUMMARY:
This pilot study examined the effect of task-oriented mobility training in three persons chronic post-stroke using a novel, wearable, mobile intention-based robotic orthosis (Tibion Bionic Leg).

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Aged 40 to 60 years
* One year status post-stroke
* Able to walk at least 10 meters
* Independence in self-care

Exclusion Criteria:

* Medically unstable
* Major cardiopulmonary deficiency
* Major depression
* Significant cognitive deficit
* Currently receiving gait training
* Younger than 40 years of age
* Older than 60 years of age
* Unable to walk at least 10 meters

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2009-06; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy N Byl, PhD, PT, Principal Investigator — University of California, San Francisco
Locations (1):
- Bakar Community Center at the University of California San Francisco, San Francisco, California, United States

REFERENCES:
- [Background] Wong CK, Bishop L, Stein J. A wearable robotic knee orthosis for gait training: a case-series of hemiparetic stroke survivors. Prosthet Orthot Int. 2012 Mar;36(1):113-20. doi: 10.1177/0309364611428235. Epub 2011 Nov 14. PMID 22082495
- See also: Tibion Bionic Technologies — http://www.tibion.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were part of the hospitals patient population.
Groups:
- Tibion Arm Baseline Assessments: Arm of the study in which enrolled post-stroke subjects undergo rehabilitative therapy with the Tibion Bionic Leg.
Period: Overall Study
Arm/Group | Tibion Arm Baseline Assessments
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: All subjects had reached plateau with conventional Bodyweight-Supported Treadmill Training (BWSTT, participated in task-oriented mobility therapy(1.5 hours, 2-4 times per week for 4 weeks) with Robotic Leg Orthosis (RLO) under the supervision of a physical therapist.
Arm/Group | All Participants
Number analyzed (Participants) | 3
Age Continuous [Median (Full Range); unit: Years] | 50 [40 to 60]
Sex: Female, Male [Count of Participants; unit: Participants] — The Baseline measurement is to specify the gender of each participant.
  Participants
    Female | 2
    Male | 1
Lower Left Extremity Strength [Median (Full Range); unit: Pounds-Force] — The strength of the left lower extremity during active extension in pounds-force (lbf).
  Pounds-Force | 105 [90 to 169]
Right Lower Extremity Strength [Median (Full Range); unit: Pounds-Force] — The strength of the right lower extremity during active extension in pounds-force (lbf).
  Pounds-Force | 105 [97 to 138]
Resting Extensor Tone (Modified Ashworth Scale) [Median (Full Range); unit: Units on a Scale] — The Modified Ashworth Scale (MAS) measures muscle hypertonia, with increasing scores signifying greater resting tone of muscle groups. Scores: 0 - No tone, 1 - Slight tone, with by a catch and release or by minimal resistance at the end of the range of motion, 1+ - Slight tone, manifested by a catch, followed by minimal resistance through less than half of the ROM, 2 - Marked increase in tone through most of ROM, but affected limb(s) easily moved, 3 - Considerable tone, passive movement difficult, 4 - Affected limb(s) rigid in flexion or extension
  Units on a Scale
    Mean Ankle Score | 2 [1 to 4]
    Mean Knee Score | 3 [1 to 4]

OUTCOME MEASURES:

1. Secondary Outcome: 6 Minute Walk Test (6 MWT)
Description: The total distance walked by the patient, in meters, as obtained by the Six (6) Minute Walk Test (6 MWT). The 6 MWT is performed over level ground, using any walking aids (canes, walkers, etc.) the patient requires for comfortable walking.
Time Frame: Baseline (prior to training); at conclusion of 4 week training regimen (1.5 hours/session with 2 to 4 sessions per week); and 1 Month post-training regimen.
Population: Three (3) Subjects all of whom had a plateaued with conventional Bodyweight-Supported Treadmill Training (BWSTT) participated in task-oriented mobility therapy (1.5 hours, 2-4 times per week for 4 weeks) with the Tibion Bionic Leg under the supervision of a physical therapist.
Measure: Number; unit: Meters
Groups:
- Patient 1; Patient 2; Patient 3: Six Minute Walk Test (meters)
Arm/Group | Patient 1 | Patient 2 | Patient 3
Number analyzed (Participants) | 1 | 1 | 1
Meters
  Baseline | 170 | 93 | 271
  End of Training | 207 | 140 | 300
  1 Month Post-Training | 250 | 123 | 285

2. Secondary Outcome: Timed Up and Go (TUG) Test
Description: The time, in seconds, for the patient to rise from sitting in a standard arm chair, walk 3 meters, turn around, walk back to the chair, and sit down. This evaluation is called the Timed Up and Go test (TUG). The patient may wear their usual footwear and use any aids (canes, walkers, etc.) they typically employ for comfortable walking.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number; unit: Seconds
Groups:
- Patient 1; Patient 2; Patient 3: Timed Up and Go Test (seconds)
Arm/Group | Patient 1 | Patient 2 | Patient 3
Number analyzed (Participants) | 1 | 1 | 1
Seconds
  Baseline | 21.4 | 21.4 | 9.14
  End of Training | 14.5 | 23.3 | 8.94
  1 Month Post-Training | 12.4 | 24.0 | 10.1

3. Secondary Outcome: Five Times Sit to Stand Test (5 x STS)
Description: The time, in seconds, for the patient to rise from a seated to full standing position and return to sitting five times in rapid succession. This evaluation is called the Five Times Sit to Stand Test (5 x STS)
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number; unit: Seconds
Groups:
- Patient 1; Patient 2; Patient 3: Five Times Sit to Stand Test (seconds)
Arm/Group | Patient 1 | Patient 2 | Patient 3
Number analyzed (Participants) | 3 | 3 | 3
Seconds
  Baseline | 12.1 | 12.4 | 11.4
  End of Training | 10.5 | 13.0 | 12.2
  1 Month Post-Training | 11.1 | 13.2 | 10.1

4. Secondary Outcome: Step Length
Description: The length of the patient's average step, in meters, as measured during comfortable walking.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number; unit: Meters
Groups:
- Patient 1; Patient 2; Patient 3: Step Length (meters)
Arm/Group | Patient 1 | Patient 2 | Patient 3
Number analyzed (Participants) | 1 | 1 | 1
Meters
  Baseline | 0.49 | 0.29 | 0.54
  End of Training | 0.56 | 0.40 | 0.59
  1 Month Post-Training | 0.59 | 0.39 | 0.60

5. Primary Outcome: Ambulation Speed
Description: Ambulation speed, in meters per second, as obtained by the Ten (10) Meter Walk Test (10 MWT). The 10 MWT measures the time required to walk 10 meters at the subject's comfortable walking pace.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number; unit: meters per second (m/s)
Groups:
- Patient 1; Patient 2; Patient 3: Ambulation speed (meters/second)
Arm/Group | Patient 1 | Patient 2 | Patient 3
Number analyzed (Participants) | 1 | 1 | 1
meters per second (m/s)
  Baseline | 0.60 | 0.29 | 0.83
  End of Training | 0.81 | 0.43 | 1.03
  1 Month Post-Training | 0.95 | 0.45 | 1.14

ADVERSE EVENTS:
Arm/Group | Tibion Arm Baseline Assessments
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 0/3

LIMITATIONS AND CAVEATS:
These results are from a small group (n of 3) of patients and should not be assumed to be consistent across all populations. Furthermore, the inherent subjective variability of patient response in physical therapy interventions should be considered.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No